CLINICAL TRIAL: NCT06343636
Title: A Phase 1, First-in-human, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study in Healthy Adults and Open-label Single Dose Study in Patients With Alzheimer's Disease to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VG-3927
Brief Title: A Phase 1 Study of VG-3927 in Healthy Adults and Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigil Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: VG3927-02.101
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single and Multiple Ascending Dose (Experimental): Ascending single doses and multiple doses for healthy volunteers.
  Interventions: Drug: VG-3927
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo
- Alzheimer's Disease (Experimental): Single Dose Open-label
  Interventions: Drug: VG-3927

INTERVENTIONS:
Drug: VG-3927 — Dose Escalation
  Arms: Single and Multiple Ascending Dose
Drug: Placebo — Dose Escalation
  Arms: Placebo
Drug: VG-3927 — One Dose Level
  Arms: Alzheimer's Disease

SUMMARY:
A Phase 1, First-in-human, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study in Healthy Adults and Open-label Single Dose Study in Patients with Alzheimer's Disease to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VG-3927.

ELIGIBILITY:
Inclusion Criteria:

* The participant is deemed healthy by the principal investigator, as determined by prestudy medical evaluation
* The participant voluntarily agrees to participate in this study and signs an institutional review board approved informed consent

Exclusion Criteria:

* The participant has any concurrent disease or condition that, in the opinion of the principal investigator, would make the participant unsuitable for participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 28 days post last dose
  To evaluate the safety and tolerability of VG-3927

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - K2 Medical Research, Maitland, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
- Nucleus Network, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No